CLINICAL TRIAL: NCT04063228
Title: High Level Mobility Training in Ambulatory Patients With Acquired Non-progressive Central Neurological Injury
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of resources
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 17-00695
Record Dates: First submitted 2019-08-19; First posted 2019-08-21 (Actual); Last update posted 2020-08-11 (Actual); Status verified 2020-08

CONDITIONS: Neurological Injury
Keywords: non-progressive central neurological injury
MeSH Terms: conditions — Trauma, Nervous System

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of care (Active Comparator)
  Interventions: Other: Simple Skill Group
- Simple Skill Group (Active Comparator)
  Interventions: Other: Complex Skill Group

INTERVENTIONS:
Other: Simple Skill Group — will practice the following skills as needed: bed mobility, transfer, walking, and stairs.
  Arms: Standard of care
Other: Complex Skill Group — The program will consist of interventions at the impairments level with an emphasis on core strengthening, functional lower extremity strengthening, balance and endurance training, and at the skill acquisition level. Participants will learn pre-running skills (walking, stairs with handrail, walking backward, walking over obstacles, walking on toes, stairs without handrail, bounding), running skills (force generation in vertical plane: hopping, alternate hopping, running in place in gravity minimized position and against gravity; force generation in horizontal plane: bounding, alternate bounding, open chain movement for swing phase, running) and post running skills (running forward, backward, sideways, skipping, hopping).
  Arms: Simple Skill Group

SUMMARY:
Brain injuries are a significant cause of loss of movement. It has been shown that physical therapy can help patients to regain movements. The purpose of this study is to see if it is possible to perform a new exercise program that will help patients regain movement. This new exercise program will involve practicing walking, stairs, jumping and running. Participation in this study will involve physical therapy 1 to 2 times a week for 12 visits over 6 to 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Referred to physical therapy with an Acquired Non-Progressive Central Neurological Injury (traumatic brain injury, stroke, brain tumor, spinal cord injury) for 3 months or more
* capacity to consent
* ability to read and write English at the sixth grade level
* able to walk twenty meter without physical assistance or an assistive device, however they can use a brace.
* self-selected gait speed of 0.6 m/s or greater when performing 10 meter walk test.

Exclusion Criteria:

* Adults subjects diagnosed with a progressive central or peripheral neurological disorder or an acute non progressive central neurological disorder (less than 3 months)
* Subjects who require physical assistance or an assistive device to walk twenty meters or demonstrate self-selected gait speed less than 0.6 m/s
* Subjects who are already able to run independently in the community
* Participants who are unable to complete the 12 physical therapy visits at prescribed skill level as established by protocol
* Participants who reports >4/10 on NPRS with lower extremity weight bearing.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2019-06-17 (Actual); Primary Completion 2020-06-01 (Actual); Study Completion 2020-06-01 (Actual)

PRIMARY OUTCOMES:
Recruitment Feasibility | 2 Years
  measured by the number of individuals who consent to participate.
Training feasibility | 2 Years
  Measured by the number of sessions attended by each participant.

CONTACTS AND LOCATIONS:
Overall Officials: Estelle Gallo, MD, Principal Investigator — New York Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States